CLINICAL TRIAL: NCT00683670
Title: Mature Dendritic Cell Vaccination Against gp100 in Patients With Advanced Melanoma
Brief Title: Dendritic Cells (White Blood Cells) Vaccination for Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0652 / 826850
Record Dates: First submitted 2008-05-19; First posted 2008-05-23 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dendritic Cell Vaccine (First Group) (Experimental): Blood mononuclear cells will be collected for vaccine production through apheresis. Patients will be given cyclophosphamide 300mg/m2 IV 3 days prior to vaccine dose #1 in order to deplete regulatory T cells. Patients will receive mature DC for each dose of vaccine and will receive autologous dendritic cells. The DC vaccine will be given intravenously every 3 weeks for a total of 6 doses. Peripheral blood will be taken weekly to monitor the immune response. Apheresis is repeated after vaccine dose #3 and dose #6 in order to collect PBMC for immune monitoring. Patients with stable disease or better after 6 doses will be eligible to receive additional vaccinations as maintenance therapy every 2 months until progression.
  Interventions: Drug: cyclophosphamide; Biological: Mature dendritic cell vaccine
- Dendritic Cell Vaccine (Second Group) (Experimental): Blood mononuclear cells will be collected for vaccine production through apheresis. Patients will be given cyclophosphamide 300mg/m2 IV 3 days prior to vaccine dose #1 in order to deplete regulatory T cells. Patients will receive mature DC for each dose of vaccine and will receive autologous dendritic cells. The DC vaccine will be given intravenously every 3 weeks for a total of 6 doses. Peripheral blood will be taken weekly to monitor the immune response. Apheresis is repeated after vaccine dose #3 and dose #6 in order to collect PBMC for immune monitoring. Patients with stable disease or better after 6 doses will be eligible to receive additional vaccinations as maintenance therapy every 2 months until progression.
  Interventions: Drug: cyclophosphamide; Biological: Mature dendritic cell vaccine
- Dendritic Cell Vaccine (Third Group) (Experimental): Blood mononuclear cells will be collected for vaccine production through apheresis. Patients will be given cyclophosphamide 300mg/m2 IV 3 days prior to vaccine dose #1 in order to deplete regulatory T cells. Patients will receive mature DC for each dose of vaccine and will receive autologous dendritic cells. The DC vaccine will be given intravenously every 6 weeks for a total of 3 doses. Peripheral blood will be taken weekly to monitor the immune response. Apheresis is repeated after vaccine dose #3 in order to collect PBMC for immune monitoring.
  Interventions: Drug: cyclophosphamide; Biological: Mature dendritic cell vaccine

INTERVENTIONS:
Drug: cyclophosphamide
  Other Names: Cytoxan
Biological: Mature dendritic cell vaccine

SUMMARY:
The purpose of this study is to investigate a method of using dendritic cells (a kind of white blood cell) as a vaccine to stimulate your own immune system to react to your melanoma cells.

DETAILED DESCRIPTION:
Eligible patients that provide written informed consent will undergo apheresis to collect blood mononuclear cells for vaccine production. All patients will be given cyclophosphamide 300mg/m2 IV three days prior to vaccine dose #1 in order to deplete regulatory T cells. All patients will receive mature DC for each dose of vaccine. For each dose all patients will receive autologous dendritic cells pulsed with 2 gp100 melanoma peptides (G209-2M and G280-9V) plus up to an additional 10 unique melanoma tumor-specific peptides. All patients will receive booster doses with mature DC. The DC vaccine will be given intravenously every three weeks for a total of six vaccine doses. Peripheral blood (16 ml) will be taken weekly to monitor the immune response to each peptide by tetramer assay. Apheresis is repeated after vaccine dose #3 and dose #6 in order to collect PBMC for immune monitoring. Restaging is performed after three and six vaccine doses. Patients with stable disease or better (partial response/complete response) after six doses will be eligible to receive additional vaccinations as maintenance therapy every 2 months until progression.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable stage III and stage IV M1a/M1b/M1c melanoma including patients with uveal melanoma
* Age ≥ 18 years
* Life expectancy ≥ 4 months
* ECOG performance status 0-2
* At least 28 days from prior treatment (including adjuvant interferon) except in cases of a BRAF inhibitor (such as vemurafenib); concurrent treatment with a BRAF inhibitor +/- MEK inhibitor is permitted
* Required initial laboratory values (submitted within 14 days prior to registration):

  * WBC >3,000/mm3
  * Hg ≥ 9.0 gm/dl
  * Platelets >75,000/mm3
  * Serum Bilirubin < 2.0 mg/dl
  * Serum Creatinine < 2.0 mg/dl
* Sexually active women of childbearing potential must use effective birth control during the trial and for at least two months following the trial, and sexually active men must be willing to avoid fathering a new child while receiving therapy.

Exclusion Criteria:

* Prior treatment with more than one line of cytotoxic chemotherapy; prior treatment with one line of cytotoxic chemotherapy is permitted. Prior treatment with targeted therapy (such as ipilumumab, anti-PD1, and BRAF inhibitor) is permitted.
* Active untreated CNS metastasis
* Active infection
* Prior malignancy (except non-melanoma skin cancer) within 3 years
* Pregnant or nursing
* Concurrent treatment with corticosteroids; local (inhaled or topical) steroids are permitted.
* Inability to provide adequate informed consent
* Known allergy to eggs
* Prior history or uveitis or autoimmune inflammatory eye disease.
* Known positivity for hepatitis BsAg, hepatitis C antibody, or HIV antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Immunological response based on measuring increased numbers of peptide specific CD8+ T cells as calculated by the tetramer assay. | Through completion of treatment
  * Starting on Day 0, two tubes will be drawn weekly until Day 64. Thereafter, two tubes will be drawn every 21 days until Day 190. For patients receiving maintenance treatment, blood is drawn every month.
  * Data are presented as the percentage of CD8+ T cells positive for tetramer binding based on gating variables set using the iMASC reagent kit (Beckman Coulter).
Safety and tolerability of the mature dendritic cell vaccine as measured by adverse events | 30 days after end of treatment
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for all toxicity reporting.

SECONDARY OUTCOMES:
Time to progression | Through completion of treatment or until progressive disease
Regulatory T cell depletion after cyclophosphamide administration. | Day -3 (72 hours prior to vaccine dose 1)
  Regulatory T cells (Treg) are defined as CD4+CD25+foxP3+ (triple positive) cells. At the indicated time points, the percentage of Treg cells is determined by 3 color flow cytometry. The depletion of Treg is defined as follows [Treg baseline - Treg nadir/ Treg baseline x 100= % depletion].
Safety and side effect profile of mDC administered to patients given after a single dose of cyclophosphamide. | Day 0 (prior to vaccine dose 1)
Clinical response rate using RECIST criteria | After third vaccine, sixth vaccine, and then every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerald P. Linette, M.D., Ph.D., Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal, A., T. Murray, E. Ward, A. Samuels, R.C. Tiwari, A. Ghafoor, E.J. Feuer, and M.J. Thun. 2007. Cancer statistics, 2007. CA Cancer J Clin 57:42-59.
- [Background] Lotze, M.T., R.M. Dallal, J.M. Kirkwood, and J.C. Flickinger. 2001. Cutaneous Melanoma. In Cancer:Principles and Practice of Oncology. V.T. DeVita, S. Hellman, and S.A. Rosenberg, editors. Lippincott, Williams, & Wilkins, Philadelphia. 2012-2069.
- [Background] Eggermont AM, Kirkwood JM. Re-evaluating the role of dacarbazine in metastatic melanoma: what have we learned in 30 years? Eur J Cancer. 2004 Aug;40(12):1825-36. doi: 10.1016/j.ejca.2004.04.030. PMID 15288283
- [Background] Queirolo P, Acquati M, Kirkwood JM, Eggermont AM, Rocca A, Testori A. Update: current management issues in malignant melanoma. Melanoma Res. 2005 Oct;15(5):319-24. doi: 10.1097/00008390-200510000-00001. PMID 16179860
- [Background] Serrone L, Zeuli M, Sega FM, Cognetti F. Dacarbazine-based chemotherapy for metastatic melanoma: thirty-year experience overview. J Exp Clin Cancer Res. 2000 Mar;19(1):21-34. PMID 10840932
- [Background] Huncharek M, Caubet JF, McGarry R. Single-agent DTIC versus combination chemotherapy with or without immunotherapy in metastatic melanoma: a meta-analysis of 3273 patients from 20 randomized trials. Melanoma Res. 2001 Feb;11(1):75-81. doi: 10.1097/00008390-200102000-00009. PMID 11254118
- [Background] Chapman PB, Einhorn LH, Meyers ML, Saxman S, Destro AN, Panageas KS, Begg CB, Agarwala SS, Schuchter LM, Ernstoff MS, Houghton AN, Kirkwood JM. Phase III multicenter randomized trial of the Dartmouth regimen versus dacarbazine in patients with metastatic melanoma. J Clin Oncol. 1999 Sep;17(9):2745-51. doi: 10.1200/JCO.1999.17.9.2745. PMID 10561349
- [Background] Ernsdorf MS, C.T., and L Titus-Ernsdorf. 2003. Update: Medical therapy for cutaneous melanoma. ASCO Educational Book 39:198-207.
- [Background] Atkins MB, Lotze MT, Dutcher JP, Fisher RI, Weiss G, Margolin K, Abrams J, Sznol M, Parkinson D, Hawkins M, Paradise C, Kunkel L, Rosenberg SA. High-dose recombinant interleukin 2 therapy for patients with metastatic melanoma: analysis of 270 patients treated between 1985 and 1993. J Clin Oncol. 1999 Jul;17(7):2105-16. doi: 10.1200/JCO.1999.17.7.2105. PMID 10561265
- [Background] Morton DL, Eilber FR, Joseph WL, Wood WC, Trahan E, Ketcham AS. Immunological factors in human sarcomas and melanomas: a rational basis for immunotherapy. Ann Surg. 1970 Oct;172(4):740-9. doi: 10.1097/00000658-197010000-00018. No abstract available. PMID 5272336
- [Background] Golub SH, Morton DL. Sensitisation of lymphocytes in vitro against human melanoma-associated antigens. Nature. 1974 Sep 13;251(5471):161-3. doi: 10.1038/251161a0. No abstract available. PMID 4421563
- [Background] Waldmann TA. Effective cancer therapy through immunomodulation. Annu Rev Med. 2006;57:65-81. doi: 10.1146/annurev.med.56.082103.104549. PMID 16409137
- [Background] Kawakami Y, Eliyahu S, Jennings C, Sakaguchi K, Kang X, Southwood S, Robbins PF, Sette A, Appella E, Rosenberg SA. Recognition of multiple epitopes in the human melanoma antigen gp100 by tumor-infiltrating T lymphocytes associated with in vivo tumor regression. J Immunol. 1995 Apr 15;154(8):3961-8. PMID 7706734
- [Background] Kawakami Y, Robbins PF, Wang RF, Parkhurst M, Kang X, Rosenberg SA. The use of melanosomal proteins in the immunotherapy of melanoma. J Immunother. 1998 Jul;21(4):237-46. doi: 10.1097/00002371-199807000-00001. PMID 9672845
- [Background] van der Bruggen P, Traversari C, Chomez P, Lurquin C, De Plaen E, Van den Eynde B, Knuth A, Boon T. A gene encoding an antigen recognized by cytolytic T lymphocytes on a human melanoma. Science. 1991 Dec 13;254(5038):1643-7. doi: 10.1126/science.1840703.
- [Background] Marincola FM, Hijazi YM, Fetsch P, Salgaller ML, Rivoltini L, Cormier J, Simonis TB, Duray PH, Herlyn M, Kawakami Y, Rosenberg SA. Analysis of expression of the melanoma-associated antigens MART-1 and gp100 in metastatic melanoma cell lines and in in situ lesions. J Immunother Emphasis Tumor Immunol. 1996 May;19(3):192-205. doi: 10.1097/00002371-199605000-00004. PMID 8811494
- [Background] Mocellin S, Mandruzzato S, Bronte V, Lise M, Nitti D. Part I: Vaccines for solid tumours. Lancet Oncol. 2004 Nov;5(11):681-9. doi: 10.1016/S1470-2045(04)01610-9. PMID 15522656
- [Background] Parmiani G, Castelli C, Santinami M, Rivoltini L. Melanoma immunology: past, present and future. Curr Opin Oncol. 2007 Mar;19(2):121-7. doi: 10.1097/CCO.0b013e32801497d7. PMID 17272984
- [Background] Bakker AB, Schreurs MW, de Boer AJ, Kawakami Y, Rosenberg SA, Adema GJ, Figdor CG. Melanocyte lineage-specific antigen gp100 is recognized by melanoma-derived tumor-infiltrating lymphocytes. J Exp Med. 1994 Mar 1;179(3):1005-9. doi: 10.1084/jem.179.3.1005. PMID 8113668
- [Background] Cox AL, Skipper J, Chen Y, Henderson RA, Darrow TL, Shabanowitz J, Engelhard VH, Hunt DF, Slingluff CL Jr. Identification of a peptide recognized by five melanoma-specific human cytotoxic T cell lines. Science. 1994 Apr 29;264(5159):716-9. doi: 10.1126/science.7513441.
- [Background] Skipper JC, Gulden PH, Hendrickson RC, Harthun N, Caldwell JA, Shabanowitz J, Engelhard VH, Hunt DF, Slingluff CL Jr. Mass-spectrometric evaluation of HLA-A*0201-associated peptides identifies dominant naturally processed forms of CTL epitopes from MART-1 and gp100. Int J Cancer. 1999 Aug 27;82(5):669-77. doi: 10.1002/(sici)1097-0215(19990827)82:53.0.co;2-#. PMID 10417764
- [Background] Salgaller ML, Marincola FM, Cormier JN, Rosenberg SA. Immunization against epitopes in the human melanoma antigen gp100 following patient immunization with synthetic peptides. Cancer Res. 1996 Oct 15;56(20):4749-57. PMID 8840994
- [Background] Rosenberg SA, Yang JC, Schwartzentruber DJ, Hwu P, Marincola FM, Topalian SL, Restifo NP, Dudley ME, Schwarz SL, Spiess PJ, Wunderlich JR, Parkhurst MR, Kawakami Y, Seipp CA, Einhorn JH, White DE. Immunologic and therapeutic evaluation of a synthetic peptide vaccine for the treatment of patients with metastatic melanoma. Nat Med. 1998 Mar;4(3):321-7. doi: 10.1038/nm0398-321. PMID 9500606
- [Background] Linette GP, Zhang D, Hodi FS, Jonasch EP, Longerich S, Stowell CP, Webb IJ, Daley H, Soiffer RJ, Cheung AM, Eapen SG, Fee SV, Rubin KM, Sober AJ, Haluska FG. Immunization using autologous dendritic cells pulsed with the melanoma-associated antigen gp100-derived G280-9V peptide elicits CD8+ immunity. Clin Cancer Res. 2005 Nov 1;11(21):7692-9. doi: 10.1158/1078-0432.CCR-05-1198. PMID 16278389
- [Background] Yee C, Savage PA, Lee PP, Davis MM, Greenberg PD. Isolation of high avidity melanoma-reactive CTL from heterogeneous populations using peptide-MHC tetramers. J Immunol. 1999 Feb 15;162(4):2227-34. PMID 9973498
- [Background] Skipper JC, Kittlesen DJ, Hendrickson RC, Deacon DD, Harthun NL, Wagner SN, Hunt DF, Engelhard VH, Slingluff CL Jr. Shared epitopes for HLA-A3-restricted melanoma-reactive human CTL include a naturally processed epitope from Pmel-17/gp100. J Immunol. 1996 Dec 1;157(11):5027-33. PMID 8943411
- [Background] Mellman I, Steinman RM. Dendritic cells: specialized and regulated antigen processing machines. Cell. 2001 Aug 10;106(3):255-8. doi: 10.1016/s0092-8674(01)00449-4. No abstract available. PMID 11509172
- [Background] Banchereau J, Schuler-Thurner B, Palucka AK, Schuler G. Dendritic cells as vectors for therapy. Cell. 2001 Aug 10;106(3):271-4. doi: 10.1016/s0092-8674(01)00448-2. No abstract available. PMID 11509176
- [Background] Nestle FO, Alijagic S, Gilliet M, Sun Y, Grabbe S, Dummer R, Burg G, Schadendorf D. Vaccination of melanoma patients with peptide- or tumor lysate-pulsed dendritic cells. Nat Med. 1998 Mar;4(3):328-32. doi: 10.1038/nm0398-328. PMID 9500607
- [Background] Thurner B, Haendle I, Roder C, Dieckmann D, Keikavoussi P, Jonuleit H, Bender A, Maczek C, Schreiner D, von den Driesch P, Brocker EB, Steinman RM, Enk A, Kampgen E, Schuler G. Vaccination with mage-3A1 peptide-pulsed mature, monocyte-derived dendritic cells expands specific cytotoxic T cells and induces regression of some metastases in advanced stage IV melanoma. J Exp Med. 1999 Dec 6;190(11):1669-78. doi: 10.1084/jem.190.11.1669. PMID 10587357
- [Background] Banchereau J, Palucka AK, Dhodapkar M, Burkeholder S, Taquet N, Rolland A, Taquet S, Coquery S, Wittkowski KM, Bhardwaj N, Pineiro L, Steinman R, Fay J. Immune and clinical responses in patients with metastatic melanoma to CD34(+) progenitor-derived dendritic cell vaccine. Cancer Res. 2001 Sep 1;61(17):6451-8. PMID 11522640
- [Background] Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. doi: 10.1038/nm1039. PMID 15122249
- [Background] Ingram SB, O'Rourke MG. DC therapy for metastatic melanoma. Cytotherapy. 2004;6(2):148-53. doi: 10.1080/14653240410005627. No abstract available. PMID 15203991
- [Background] Randolph DA, Fathman CG. Cd4+Cd25+ regulatory T cells and their therapeutic potential. Annu Rev Med. 2006;57:381-402. doi: 10.1146/annurev.med.57.121304.131337. PMID 16409156
- [Background] Roncador G, Brown PJ, Maestre L, Hue S, Martinez-Torrecuadrada JL, Ling KL, Pratap S, Toms C, Fox BC, Cerundolo V, Powrie F, Banham AH. Analysis of FOXP3 protein expression in human CD4+CD25+ regulatory T cells at the single-cell level. Eur J Immunol. 2005 Jun;35(6):1681-91. doi: 10.1002/eji.200526189. PMID 15902688
- [Background] Antony PA, Restifo NP. CD4+CD25+ T regulatory cells, immunotherapy of cancer, and interleukin-2. J Immunother. 2005 Mar-Apr;28(2):120-8. doi: 10.1097/01.cji.0000155049.26787.45. PMID 15725955
- [Background] Lutsiak ME, Semnani RT, De Pascalis R, Kashmiri SV, Schlom J, Sabzevari H. Inhibition of CD4(+)25+ T regulatory cell function implicated in enhanced immune response by low-dose cyclophosphamide. Blood. 2005 Apr 1;105(7):2862-8. doi: 10.1182/blood-2004-06-2410. Epub 2004 Dec 9. PMID 15591121
- [Background] Ko K, Yamazaki S, Nakamura K, Nishioka T, Hirota K, Yamaguchi T, Shimizu J, Nomura T, Chiba T, Sakaguchi S. Treatment of advanced tumors with agonistic anti-GITR mAb and its effects on tumor-infiltrating Foxp3+CD25+CD4+ regulatory T cells. J Exp Med. 2005 Oct 3;202(7):885-91. doi: 10.1084/jem.20050940. Epub 2005 Sep 26. PMID 16186187
- [Background] Nomura T, Sakaguchi S. Naturally arising CD25+CD4+ regulatory T cells in tumor immunity. Curr Top Microbiol Immunol. 2005;293:287-302. doi: 10.1007/3-540-27702-1_13. PMID 15981485
- [Background] Sakaguchi S, Sakaguchi N. Regulatory T cells in immunologic self-tolerance and autoimmune disease. Int Rev Immunol. 2005 May-Aug;24(3-4):211-26. doi: 10.1080/08830180590934976. PMID 16036375
- [Background] Bass KK, Mastrangelo MJ. Immunopotentiation with low-dose cyclophosphamide in the active specific immunotherapy of cancer. Cancer Immunol Immunother. 1998 Sep;47(1):1-12. doi: 10.1007/s002620050498. PMID 9755873
- [Background] Hoon DS, Foshag LJ, Nizze AS, Bohman R, Morton DL. Suppressor cell activity in a randomized trial of patients receiving active specific immunotherapy with melanoma cell vaccine and low dosages of cyclophosphamide. Cancer Res. 1990 Sep 1;50(17):5358-64. PMID 2143687
- [Background] Miles DW, Towlson KE, Graham R, Reddish M, Longenecker BM, Taylor-Papadimitriou J, Rubens RD. A randomised phase II study of sialyl-Tn and DETOX-B adjuvant with or without cyclophosphamide pretreatment for the active specific immunotherapy of breast cancer. Br J Cancer. 1996 Oct;74(8):1292-6. doi: 10.1038/bjc.1996.532. PMID 8883420
- [Background] Steinman RM, Pope M. Exploiting dendritic cells to improve vaccine efficacy. J Clin Invest. 2002 Jun;109(12):1519-26. doi: 10.1172/JCI15962. No abstract available. PMID 12070296
- [Background] Belardelli F, Ferrantini M, Parmiani G, Schlom J, Garaci E. International meeting on cancer vaccines: how can we enhance efficacy of therapeutic vaccines? Cancer Res. 2004 Sep 15;64(18):6827-30. doi: 10.1158/0008-5472.CAN-04-2048. PMID 15375003
- [Background] Lin AM, Hershberg RM, Small EJ. Immunotherapy for prostate cancer using prostatic acid phosphatase loaded antigen presenting cells. Urol Oncol. 2006 Sep-Oct;24(5):434-41. doi: 10.1016/j.urolonc.2005.08.010. PMID 16962496
- [Background] Pulendran B, Palucka K, Banchereau J. Sensing pathogens and tuning immune responses. Science. 2001 Jul 13;293(5528):253-6. doi: 10.1126/science.1062060. PMID 11452116
- [Background] Moss P, Khan N. CD8(+) T-cell immunity to cytomegalovirus. Hum Immunol. 2004 May;65(5):456-64. doi: 10.1016/j.humimm.2004.02.014. PMID 15172445
- [Background] Keilholz U, Weber J, Finke JH, Gabrilovich DI, Kast WM, Disis ML, Kirkwood JM, Scheibenbogen C, Schlom J, Maino VC, Lyerly HK, Lee PP, Storkus W, Marincola F, Worobec A, Atkins MB. Immunologic monitoring of cancer vaccine therapy: results of a workshop sponsored by the Society for Biological Therapy. J Immunother. 2002 Mar-Apr;25(2):97-138. doi: 10.1097/00002371-200203000-00001. PMID 12074049
- [Background] Grover A, Kim GJ, Lizee G, Tschoi M, Wang G, Wunderlich JR, Rosenberg SA, Hwang ST, Hwu P. Intralymphatic dendritic cell vaccination induces tumor antigen-specific, skin-homing T lymphocytes. Clin Cancer Res. 2006 Oct 1;12(19):5801-8. doi: 10.1158/1078-0432.CCR-05-2421. PMID 17020987
- [Background] Torabian S, Kashani-Sabet M. Biomarkers for melanoma. Curr Opin Oncol. 2005 Mar;17(2):167-71. doi: 10.1097/01.cco.0000154039.07466.5d. PMID 15725923
- [Derived] Carreno BM, Magrini V, Becker-Hapak M, Kaabinejadian S, Hundal J, Petti AA, Ly A, Lie WR, Hildebrand WH, Mardis ER, Linette GP. Cancer immunotherapy. A dendritic cell vaccine increases the breadth and diversity of melanoma neoantigen-specific T cells. Science. 2015 May 15;348(6236):803-8. doi: 10.1126/science.aaa3828. Epub 2015 Apr 2. PMID 25837513
- [Derived] Carreno BM, Becker-Hapak M, Huang A, Chan M, Alyasiry A, Lie WR, Aft RL, Cornelius LA, Trinkaus KM, Linette GP. IL-12p70-producing patient DC vaccine elicits Tc1-polarized immunity. J Clin Invest. 2013 Aug;123(8):3383-94. doi: 10.1172/JCI68395. Epub 2013 Jul 11. PMID 23867552
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu